CLINICAL TRIAL: NCT04454723
Title: Impact of Palliative Transfusions on Quality of Life in Patients With Hematological Malignancies on Hospice - A Case Series Study
Brief Title: Impact of Palliative Transfusions on Quality of Life in Patients With Blood Cancers on Hospice
Acronym: PalliaQOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OU-SCC-PalliativeQOL
Record Dates: First submitted 2020-06-12; First posted 2020-07-01 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Hematologic Malignancy
Keywords: hospice
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Platelet Transfusion; Blood Cell Count

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tranfusions and blood collection (Experimental): Patients enrolled will receive one unit each of blood and/or platelet transfusions once a week based on trigger symptoms of anemia and/or thrombocytopenia, along with blood sample collections.
  Data on patient demographics, disease, and length of hospice stay will also be collected.
  Interventions: Procedure: Blood and/or platelet transfusion; Procedure: Complete blood count (CBC) collection

INTERVENTIONS:
Procedure: Blood and/or platelet transfusion — The transfused patients will receive one unit each of blood and/or platelet transfusions once a week based on CTCAE symptom grade 2 or greater of anemia and/or thrombocytopenia.
Procedure: Complete blood count (CBC) collection — CBC will be collected from patients weekly while on this protocol.

SUMMARY:
The purpose of this pilot research study is to evaluate the effectiveness of blood and platelet transfusions in improving symptoms and quality of life of patients enrolled in hospice.

DETAILED DESCRIPTION:
This is a non-randomized pilot study to investigate the feasibility of symptom-based blood transfusion in patients with hematologic malignancies enrolling in hospice care.

The study will be a case series involving OU Medical Center (OUMC). Patients will be identified at the University of Oklahoma/Stephenson Cancer Center (OU-SCC) where investigators performing the study will consent and monitor patients. Integris Home Hospice agency will provide hospice patients with blood transfusions in those willing to participate, and the Oklahoma Blood Institute (OBI) will provide the hospice patients with palliative transfusions at home at no cost to the patient, including blood products, transfusion testing, infusions and the nursing staff.

This will be a pilot project including 20 consented patients with hematologic malignancies enrolling in hospice through Integris Home Hospice. The transfusions received will be determined by the hospice team, and will not be based on objective symptom based guidelines. Patients will have the option to either be enrolled on this clinical trial, where they may receive home based blood or platelet transfusions, or be enrolled in any other hospice of their choosing, including the other hospice that will provide home based transfusions. Information will be collected regarding symptoms, Hospice QOL scores and transfusion use, reactions, and time in hospice. Data will be collected until death.

ELIGIBILITY:
Patients >= 18 years irrespective of their race, sex and/or other medical history.

Inclusion Criteria:

* All patients >= 18 years with a primary diagnosis of acute myeloid leukemia (AML), acute lymphoblastic leukemia (ALL), chronic lymphocytic leukemia (CLL), chronic myelomonocytic leukemia (CMML), "high risk" Non-Hodgkin's Lymphoma (NHL), multiple myeloma (MM) and Myelodysplastic Syndrome (MDS) with a life expectancy of < 6 months who are transfusion dependent. Criteria for transfusion dependence is Symptom Questionnaire symptom grade 2 or higher. The Symptom Questionnaire is based on CTCAE (Common Terminology Criteria for Adverse Events) v5.0, with criteria modified for palliative care patients.
* Patients wanting to enroll in hospice.
* Availability of peripheral IV access line or patient agrees to have semi-permanent IV line placed.

Exclusion Criteria:

* Patients with > 6-month survival.
* Patients unwilling to go on hospice.
* Patients with antibodies to blood or platelets that would preclude ability to give blood/platelets without prolonged blood typing and or need for anti-HLA platelets.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-08-14 (Actual); Primary Completion 2023-08-16 (Actual); Study Completion 2023-08-17 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with improved quality of life after receiving transfusions. | 6 months
  Improved quality of life (QOL) and palliative efficacy will be evaluated by improvement of the presenting symptoms and quality of life based on CTCAE and QOL questionnaires.
Proportion of subjects with improved palliative efficacy after receiving transfusions. | 6 months
  Palliative efficacy will be evaluated by improvement of the presenting symptoms and quality of life based on CTCAE and QOL questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Holter, MD, Principal Investigator — University of Oklahoma
Locations (1):
- Stephenson Cancer Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No